CLINICAL TRIAL: NCT05827835
Title: A Study to Evaluate the Efficacy and Safety of CD7CAR-T Bridging to Allogeneic Hematopoietic Stem Cell Transplantation in Patients With Refractory or Relapsed CD7 Positive Malignant Hematologic Diseases
Brief Title: CD7 CAR-T Bridging to alloHSCT for R/R CD7+Malignant Hematologic Diseases
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2022023
Record Dates: First submitted 2023-03-30; First posted 2023-04-25 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Hematologic Diseases; Neoplasms
Keywords: allo-HSCT; CD7 CAR-T
MeSH Terms: conditions — Hematologic Diseases; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): R/R CD7+Malignant Hematologic Diseases
  Interventions: Drug: CD7 CAR-T cells injection; Other: Allogeneic hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: CD7 CAR-T cells injection — CD7 CAR T cells treat patients with refractory or relapsed CD7 positive Malignant Hematologic Diseases
Other: Allogeneic hematopoietic stem cell transplantation — In this study, Allogeneic hematopoietic stem cell transplantation is used as a bridge therapy to CD7 CAR T cells infusion to treat patients with refractory or relapsed CD7 positive Malignant Hematologic Diseases

SUMMARY:
This is a single-arm, open-label, single-center, phase I/II study. The primary objective is to evaluate the safety of CD7 CAR-T Bridging to allo-HSCT therapy for patients with CD7-positive relapsed or refractory Malignant Hematologic Diseases

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form (ICF)
* Male or female, older than 18 years (including 18 years)
* Anticipated survival time more than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* According to the National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines for Acute Lymphocytic Leukemia and Acute Myeloid Leukemia (2016. v1), patients diagnosed as CD7+ALL and AML
* Consistent with r/r CD7+acute leukemia diagnosis, including any of the following conditions
* a. No CR after standard chemotherapy
* b. The first induction reaches CR, but CR ≤ 12 months
* c. Patients with r/r CD7+acute leukemia have not responded to the first or multiple remedial treatments
* d. Multiple recurrences
* Philadelphia chromosome negative (Ph -) subjects; Or cannot tolerate tyrosine kinase inhibitor (TKI) treatment; Or Philadelphia chromosome positive (Ph+) subjects who did not respond to both TKI treatments
* Normal lung function, oxygen saturation greater than 92% without oxygen inhalation
* The blood biochemical test results are consistent with the following results
* a. (AST) and (ALT) ≤ 2.5 × (ULN)
* b. Total bilirubin ≤ 1.5 × ULN
* c. 24-hour serum creatinine clearance ≥ 30 mL/min
* d. Lipase and amylase ≤ 2 × ULN
* Fertility capable men and women of childbearing age must agree to use effective contraception starting with the signing of an informed consent form until within 2 years after the use of the study drug. Women of reproductive age include pre menopausal women and women within 2 years after menopause. The blood pregnancy test for women of reproductive age must be negative at screening

Exclusion Criteria:

* Patients with the history of epilepsy or other CNS disease
* Pregnant or breastfeeding
* Active infection with no cure
* Patients with prolonged QT interval time or severe heart disease
* Have experienced hypersensitivity or intolerance to any drug used in this study
* Patients who received anticancer chemotherapy or other drug treatment within 2 weeks before screening
* Previous malignant tumors that require treatment or have evidence of recurrence within the previous 5 years of screening
* Clinically significant central nervous system lesions such as seizures, cerebral vascular ischemia/hemorrhage, dementia, cerebellar disease, psychosis, active central nervous system involvement, or cancerous meningitis
* In the past 2 years, terminal organ damage caused by autoimmune diseases (such as Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) or the need for systematic application of immunosuppressive or other systemic disease control drugs
* Severe active viral, bacterial, or uncontrolled systemic fungal infections; Genetic bleeding/coagulation disorders, a history of non-traumatic bleeding or thromboembolism, and other diseases that may increase the risk of bleeding
* Patients who received autologous hematopoietic stem cell transplantation (ASCT) within 8 weeks before screening, or who plan to undergo ASCT during this study
* Participated in clinical trials of other drugs within 4 weeks or 5 drug half-lives (T1/2) before screening
* Any situation that the researchers believe may increase the risk of patients or interfere with the test results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2026-04-25 (Estimated); Study Completion 2027-04-25 (Estimated)

PRIMARY OUTCOMES:
Incidence and level of AE and SAE | Baseline up to 28 days after CD7 CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria

SECONDARY OUTCOMES:
CAR-T cell expression | Evaluate at 1, 2, 3, 4, 8,12,16, 20 and 24 weeks after CAR-T infusion
  CAR-T cell expression in vivo
CAR-T related cytokine expression | Evaluate at 1, 2, 3 and 4 weeks after CAR-T infusion
  CAR-T related cytokine expression
Survival Rate （SR） | Evaluate at 6, 9, and 12 months
  Survival Rate （SR）
Time-To-Progression（TTP） | Month 2,3,4,6,12,18and 24
  Time from the beginning of treatment to the progression of the disease
Progression-free survival (PFS) | Month 6,12,18and 24
  Assessment of PFS at Month 6,12,18and 24
Duration of remission,DOR | Up to 1 years after Treatment
  The time from CR/CRi and PR to disease relapsed or death due to disease progression after CAR-T infusion
Overall response rate,ORR | Evaluate at 4, 8, and 12 weeks after CAR-T infusion
  The proportion of patients with CR (complete remission) /CRi (complete remission with incomplete blood count recovery); The proportion of patients with CR (complete response) /CRi (complete response with incomplete blood cell recovery) and PR (partial response).
Clinical Benefit Rate（CBR） | Up to 24 weeks after Treatment
  ORR+MR
Disease Control Rate （DCR） | Up to 12 weeks after Treatment
  CBR+SD
Overall survival, OS | Up to 1 years after Treatment
  The time from CAR-T infusion to death due to any cause
Minimal Residual Disease | Up to 2 years after Treatment
  MRD in CR and sCR patients
Bone marrow transplantation STR | Evaluate at 4, 8,12,16 and 20 weeks after allogeneic hematopoietic stem cell transplantation
  Monitoring the status of allogeneic hematopoietic stem cell transplantation using STR-PCR

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China